CLINICAL TRIAL: NCT04487626
Title: Development and Validation of an Artificial Intelligence System for Bowel Preparation Quality Scoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Dae Kyung Sohn, Staff surgeon, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NCC2020-0159
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Colonic Disease
Keywords: artificial intelligence, deep learning, bowel preparation
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artificial Intelligence assisted Scoring Group (Experimental): Patients in this group go through colonoscopy under the AI monitoring device.
  Interventions: Device: AI

INTERVENTIONS:
Device: AI — After taking standard bowel preparation regimen, patients receive colonoscopy under the AI system device. During the withdrawal phase, bowel preparation quality is assessed by AI-associated scoring system. The withdrawal time is targeted at least 6min. Every detected polyp will be removed and obtained for pathological assessment.

SUMMARY:
The purpose of this study is to develop and validate the accuracy and reliability of an artificial intelligence(AI) system for bowel preparation quality scoring based of Boston Bowel preparation Scoring(BBPS). Then evaluate whether this AI system can help endoscopists to improve the quality of colonoscopy in clinical practice.

DETAILED DESCRIPTION:
Bowel preparation is one of the most important factors which decide the quality of colonoscopy. Adequate bowel preparation is essential to guarantee a clear vision of colonic mucosa, complete inspection of entire colon and improves the adenoma detection rates(ADRs). Therefore, the quality of bowel preparation should be evaluated accurately and objectively. However, current bowel preparation quality scales depend on memories and subjective decision of endoscopists. Recently, articifial intelligence system based on deep learning algorithm has been used widely in medical fields. But, few studies have been reported to evaluate the performance of AI system based on deep learning in bowel preparation quality scoring. This study aims to develop and train an AI system to assess bowel preparation quality using the BBPS, and validate the AI system to improve the quality of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-80 years undergoing elective colonoscopy

Exclusion Criteria:

* Patients received colon or rectal surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
accuracy of bowel preparation score | 6 months
  Bowel preparation quality was measured by BBPS. After fully washing or suctioning of colonic contents, three segments including right colon (containing cecum and ascending colon), transvers colon (containing hepatic and splenic flexures) and left colon (containing descending and sigmoid colon) were individually scored from 0 to 3. Point 0 refers to unprepared colon segment with obscured solid stool making mucosa cannot be seen; Point 1 refers to part of mucosa can be seen, but some areas are covered by staining, residual stool, and/or opaque liquid; Point 2 refers to entire mucosa is well-seen; Point 3 refers to clean colon segment without staining, fecal materials or liquids. A sub-score of each colon segment was used, ranging from minimum 0 to maximum 3. The highest score means the excellent bowel preparation. Adequate bowel preparation was defined as a total BBPS≥6 and sub-BBPS≥2 per segment.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No